CLINICAL TRIAL: NCT00660933
Title: Intravenous Iron Versus Oral Iron for Severe Postpartum Anemia Randomized Trial
Brief Title: Intravenous Iron Versus Oral Iron for Severe Postpartum Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Montse Palacio, Hospital Clínic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POSTPARTFEEV
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2005-09

CONDITIONS: Anemia; Puerperal Disorders
Keywords: postpartum anemia; intravenous iron
MeSH Terms: conditions — Anemia; Puerperal Disorders | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Group A: Administration of intravenous iron sucrose.
  Interventions: Drug: Iron sucrose
- Group B (Placebo Comparator): Group B: Administration of intravenous NaCl 0,9%.
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Iron sucrose — Iron sucrose 200 mg/day iv, (20 mg/ml) + 200 cc de NaCl 0,9%/day in 60 minutes per 2 days.
  Other Names: Venofer
  Arms: Group A
Drug: NaCl — NaCl 0,9% 200 ml /day iv in 60 minutes per 2 days
  Arms: Group B

SUMMARY:
The aim of the study is to compare the effect of intravenous versus oral iron in women with severe postpartum anemia.

DETAILED DESCRIPTION:
Postpartum anemia is commonly defined as hemoglobin levels less than 8.5 g/dl and it is usually treated with oral iron supplements. Blood transfusion is reserved to women with hemoglobin levels < 6 g/dl and/or clinical symptoms of anemia. Without treatment, the restoration of blood parameters in postpartum anemia can take approximately one month (hemoglobin levels increase to 2.8 g/dl in 30 days). Several reports have demonstrated the efficacy of intravenous iron in severe anemia in non-obstetric pathologies. However, the clinical effect of intravenous iron in patients with postpartum hemoglobin levels ranging from 6.0 to 8.0 g/dl has been not reported. There has not been evaluated its capacity to restore hemoglobin levels and to minimize clinical side-effects of anemia (sickness, weariness, depression, anxiety).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older,
2. Diagnosis of postpartum anemia within the first 48 h postpartum with an haemoglobin level equal or higher than 6 g/dL and lower than 8.0 g/dL,
3. Ability to read and understand the relevant purpose of the trial and consent obtained in accordance with specifications of the local research ethics committee.

Exclusion Criteria:

1. Clinical symptoms or suspicion of acute or chronic infection.
2. Allergic history or iron intolerance.
3. Indication of blood transfusion.
4. Non iron deficit anemia.
5. Hepatopathy.
6. Parenteral iron hypersensitivity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To evaluate if intravenous iron administration is better than oral treatment to improve hemoglobin and hematocrit parameters in women with severe postpartum anemia | 6 weeks

SECONDARY OUTCOMES:
To compare if the administration of intravenous iron supplementation is better than the oral dosage to reestablish clinical symptoms of severe anemia minimizing its side-effects (weariness, depression, anxiety) or to avoid the need for blood transfusion | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Montse Palacio, MD, PhD, Principal Investigator — Servei de Medicina Maternofetal. Institut de Ginecologia, Obstetrícia i Neonatología. Hospital Clínic. Universitat de Barcelona
Locations (1):
- Hospital Clínic of Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Perello MF, Coloma JL, Masoller N, Esteve J, Palacio M. Intravenous ferrous sucrose versus placebo in addition to oral iron therapy for the treatment of severe postpartum anaemia: a randomised controlled trial. BJOG. 2014 May;121(6):706-13. doi: 10.1111/1471-0528.12480. Epub 2014 Jan 15. PMID 24423186